CLINICAL TRIAL: NCT02600390
Title: An Open-label, Repeated-dose, Dose Escalation Study of the Safety and Effectiveness of SANGUINATE™ for the Treatment of Leg Ulcers in Adult Patients With Sickle Cell Disease
Brief Title: SANGUINATE™ in Sickle Cell Disease Associated Leg Ulcer
Acronym: LU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prolong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGSC-009
Record Dates: First submitted 2015-11-02; First posted 2015-11-09 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Leg Ulcer
Keywords: Leg Ulcer; LU; SANGUINATE; QOL; SCD; Sickle Cell Disease; Sickle Cell; Anemia; Leg Wound; Leg; Skin Lesion
MeSH Terms: conditions — Leg Ulcer; Anemia, Sickle Cell; Anemia | interventions — PEGylated carboxyhemoglobin bovine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SANGUINATE™ (4-week) (Experimental): This is an Open-label, repeated-dose study. About five patients will be observed for 3 weeks continuing on standard of care therapy (for wound cleaning and bandaging). This will be followed by a 4-week treatment period to include once weekly doses of SANGUINATE provided via two-hour IV infusion. The final week of the study will include another observation period wherein all patients will receive standard of care therapy.
  Interventions: Biological: SANGUINATE
- SANGUINATE™ (6-week) (Experimental): This is an Open-label, repeated-dose study. About five patients will be observed for 3 weeks continuing on standard of care therapy (for wound cleaning and bandaging). This will be followed by a 6-week treatment period to include once weekly doses of SANGUINATE provided via two-hour IV infusion. The final week of the study will include another observation period wherein all patients will receive standard of care therapy.
  Interventions: Biological: SANGUINATE

INTERVENTIONS:
Biological: SANGUINATE — A two-hour infusion provided once a week over a 4-week or 6-week period.

SUMMARY:
SANGUINATE™ Sickle Cell Disease associated Leg Ulcers.

DETAILED DESCRIPTION:
This is an escalating, repeated-dose, open-label Phase 2 study to test SANGUINATE (pegylated carboxyhemoglobin bovine) in patients suffering from leg ulceration associated with Sickle Cell Disease (SCD leg ulcer).

Patients will undergo consent and screening procedures at the time of presentation for leg ulcer treatment. Eligible patients will begin a 3-week Run-In Period. A total of approximately fifteen (15) patients are expected to be screened in order to achieve an enrollment target of ten (10) evaluable patients for participation in the study. Evaluable is defined as a patient receiving a minimum of three doses of investigational product. Five (5) patients (Cohort 1) will receive four (4) once-weekly 2-hour IV infusions of SANGUINATE at a dose of 320 mg/kg (8 mL). An additional five (5) patients (Cohort 2) will receive six (6) once-weekly 2-hour IV infusions of SANGUINATE also at a dose of 320 mg/kg. Each patient will be contacted by telephone approximately 24 hours after dosing to verify the safety status of the patient. One week following the Treatment Phase, patients will return to the study center for a Final Visit where safety assessments will be performed. During the Final Visit, patients will receive standard of care treatment of ulcer. All patients will receive once-weekly Standard of Care (SOC) therapy for SCD leg ulcer for the duration of the study. SOC includes dressing the wound with multi-layer, short stretch, compression bandaging. Non-adherent, medical-grade foam will be used as the wound contact layer and primary dressing.

ELIGIBILITY:
Inclusion Criteria:

* Properly consented patients suffering from Sickle Cell Disease (Hb-SS or Hb- Sβ° genotype) associated Leg ulcer.
* Presence of leg ulcer for at least 4 weeks
* Venous Clinical Severity Score of moderate to severe (defined as ≥12)
* Leg ulcer below the knee

Exclusion Criteria:

* Patient presenting with a clinically & laboratory confirmed bacterial, fungal or acid fast organisms
* Patient has a recent acute complication of Sickle Cell Disease (e.g., pain crisis within 7 days, or acute chest syndrome within 21 days)
* Patient is planning to be pregnant, is pregnant, or is breast-feeding
* Presence of moderate to severe renal insufficiency (CrCl < 30 mL/min) or chronic kidney disease, or of moderate to severe hepatic insufficiency (Child-Pugh class B or C)
* Patients with more than 3 times the upper limit of normal laboratory reference range
* Concurrent or recent prior treatment (within 90 days) with an investigational medication
* Patients currently receiving treatment with hydroxyurea must be on stable dose for at least 30 days
* Receipt of a blood transfusion within 21 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Safety of treatment as determined by changes in vital signs, electrocardiographic, biochemical, hematological, and urinalysis measures, and reported adverse events | 8 or 10 weeks
Change in Sickle Cell Disease leg ulcer wound pain scores as measured by a 10-point scale, relative to non-wound site pain scores | 8 or 10 weeks
Rate and extent of leg ulcer wound healing as measured by change in wound surface area | 8 or 10 weeks

SECONDARY OUTCOMES:
Changes in leg ulcer wound status as measured by need for debridement (type and quantity of non-viable tissue) | 8 or 10 weeks
Changes in leg ulcer wound status as measured by extent of exudate production | 8 or 10 weeks
  Change in quality of life as measured by SF-12 Health Survey (acute version) as well as other indicators of patient comfort and well-being
Changes in leg ulcer wound status as measured by type and amount of granulation tissue | 8 or 10 weeks
Changes in leg ulcer wound status as measured by overall change in leg ulcer wound appearance | 8 or 10 weeks
Change in local skin in the region of the leg ulcer as measured by skin appearance (coloration, inflammation, etc.) | 8 or 10 weeks
Change in local skin in the region of the leg ulcer as measured by skin temperature (relative to body temperature) | 8 or 10 weeks
Improvement in leg ulcer wound severity as measured by Venous Clinical Severity Score (VCSS) | 8 or 10 weeks
Change in quality of life, as measured by an SF-12 Health Survey (acute version) as well as other indicators of patient comfort and well-being | 8 or 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hemant Misra, PhD, Study Director — Prolong Pharma
Locations (2):
- General Hospital Plaza de la Salud, Santo Domingo, Dominican Republic
- Centro Hemato-Oncologico, Marbella, Panama

IPD SHARING:
Plan to Share IPD: No